CLINICAL TRIAL: NCT03010228
Title: Study Assessing the Safety, Immunogenicity and Dose Response of VLA15, A New Multivalent Recombinant OspA Vaccine Candidate Against Lyme Borreliosis, In Healthy Adults Aged Below 40 Years
Brief Title: Study Assessing the Safety, Immunogenicity and Dose Response of VLA15, A New Vaccine Candidate Against Lyme Borreliosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VLA15-101; C4601005 (Other: Alias Study Number)
Record Dates: First submitted 2016-12-21; First posted 2017-01-04 (Estimated); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Lyme Borreliosis, Nervous System
Keywords: VLA15; Lyme Borreliosis; Multivalent Recombinant OspA Vaccine
MeSH Terms: conditions — Lyme Neuroborreliosis; Lyme Disease | interventions — aluminum sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- VLA15 12 µg with Alum (Active Comparator): VLA15 12 µg (microgram) with Alum has an injection volume of 100 µl (microliter). The amount of Alum per injection is 0.05 mg (milligram).
  Interventions: Biological: VLA15 with Alum
- VLA15 12 µg w/o Alum (Active Comparator): VLA15 12 µg (microgram) without (w/o) Alum (aluminum hydroxide) has an injection volume of 100 µl (microliter).
  Interventions: Biological: VLA15 without Alum
- VLA15 48 µg with Alum (Active Comparator): VLA15 48 µg (microgram) with Alum (aluminum hydroxide) has an injection volume of 400 µl (microliter). The amount of Alum per injection is 0.2 mg (milligram).
  Interventions: Biological: VLA15 with Alum
- VLA15 48 µg w/o Alum (Active Comparator): VLA15 48 µg (microgram) without (w/o) Alum (aluminum hydroxide) has an injection volume of 400 µl (microliter).
  Interventions: Biological: VLA15 without Alum
- VLA15 90 µg with Alum (Active Comparator): VLA15 90 µg (microgram) with Alum (aluminum hydroxide) has an injection volume of 750 µl (microliter). The amount of Alum per injection is 0.375 mg (milligram).
  Interventions: Biological: VLA15 with Alum
- VLA15 90 µg w/o Alum (Active Comparator): VLA15 90 µg (microgram) without (w/o) Alum (aluminum hydroxide) has an injection volume of 750 µl (microliter).
  Interventions: Biological: VLA15 without Alum

INTERVENTIONS:
Biological: VLA15 with Alum — I.M. vaccination with a multivalent outer surface protein A (OspA) based vaccine candidate on days 0, 28 and 56; three different doses
  Arms: VLA15 12 µg with Alum; VLA15 48 µg with Alum; VLA15 90 µg with Alum
Biological: VLA15 without Alum — I.M. vaccination with a multivalent outer surface protein A (OspA) based vaccine candidate on days 0, 28 and 56; three different doses
  Arms: VLA15 12 µg w/o Alum; VLA15 48 µg w/o Alum; VLA15 90 µg w/o Alum

SUMMARY:
Observer-blind, partially randomized, multi-center dose escalation Phase I study in healthy adults below 40 years of age.

180 subjects will be enrolled in 6 treatment groups (different doses; different formulation: with/without adjuvant); vaccinations will be given I.M.(intramuscular) into the deltoid region on Days 0, 28 and 56. Study participants will be followed up until one year after first vaccination.

Booster Extension:

Subjects in the 48µg and 90µg Treatment groups who received a complete Primary immunization schedule will be included into a Booster Extension 13 months after the first immunization.

DETAILED DESCRIPTION:
This is an observer-blind, partially randomized, multi-center dose escalation Phase I study which aims to assess the safety, immunogenicity and dose response of VLA15 in healthy adults aged below 40 years.

Overall 180 subjects will be enrolled in 6 treatment groups: VLA15 12µg with and w/o (without) Alum, VLA15 48µg with and w/o Alum, VLA15 90µg with and w/o Alum.

For the first 24 subjects, the study will be open-label and subjects will not be randomized but included into a staggered dose escalation scheme for safety precaution. Thereafter, the study will be conducted observer-blind in respect to the investigators and site staff involved in clinical evaluation of subjects, subjects will be blinded as well. Remaining 156 subjects will be randomized into the 6 treatment groups. I.M. vaccinations are administered on Days 0, 28 and 56 into deltoid region of the non-dominant arm.

The study will investigate the safety and tolerability as well as immunogenicity of VLA15. The primary objective addresses safety and tolerability of the vaccine up to three months after enrollment, i.e. 84 days after first vaccination. The study includes 1 screening visit and 8 outpatient visits from day 0 through day 365. In addition, safety phone calls will be performed.

Booster Extension:

Subjects in the 48µg and 90µg dose Groups at the Belgian site, who received a complete primary immunization schedule (three vaccinations), will be included into a Booster Extension to investigate the safety and immunogenicity of a booster dose of VLA15 administered 13 months after the first immunization. An extension analysis on safety and immunogenicity will be performed after the last subject has completed the last study visit at Month 19. Additionally a M14 interim analysis on immunogenicity data will be performed, when all subjects completed Month 14.

For inclusion in the Booster Extension of this study only subjects are eligible, who were enrolled in Belgium, completed the primary immunization schedule (three vaccinations) and were randomized into 48µg or 90µg dose groups with or without alum. Subjects included in the staggered dose escalation phase will not be asked to participate in the Booster Extension for operational reasons.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults ≥18 to <40 years of age (for US healthy adults ≥ 19 years to <40 years) at the time of screening. Health status is assessed by investigator at time of screening based on medical history, physical examination, and laboratory parameters.
* Written informed consent obtained from the subject prior to any study related procedures.
* BMI ≥18.5 and <30 at Visit 0 (Screening Visit).
* Men or women; women require a negative pregnancy test at screening. Women with childbearing potential must agree to use an adequate contraception during the entire study.

Booster Extension:

* Completed Primary immunization schedule (three vaccinations)
* Randomization into 48µg or 90µg group with or without Alum
* Written informed consent for Booster Extension obtained from the subject prior to any study related procedures.
* Enrolled at study site in Belgium
* Men or women; women require a negative pregnancy test before booster vaccination. Women of childbearing potential must agree to use an adequate contraception during the entire study.

Exclusion Criteria:

* Pathological findings in any of the investigations (i.e. medical history, physical examination) as deemed clinically relevant by the investigator or any abnormal laboratory parameter of hematology, clinical chemistry, coagulation, RF (Rheumatoid Factor) or ACPA (Anti-citrullinated protein antibodies) at the Screening Visit.
* Medical history of severe cardiovascular, respiratory (including asthma), metabolic, neurological, hepatic, rheumatic, hematological, gastrointestinal, renal disorders.
* Medical history of or current musculoskeletal disorders as deemed clinically relevant by the investigator, arthritis or chronic musculoskeletal pain.
* Previous vaccination against Lyme borreliosis with any (investigational) vaccine.
* Use of any other investigational or non-registered medicinal product within 30 days prior to VLA15 vaccination at Visit 1 (Day 0) and throughout the entire study period.
* Chronic illness related to Lyme borreliosis (LB), a history of or active symptomatic LB as suspected or diagnosed by a physician. Subjects with a positive serology test result for Borrelia burgdorferi sensu lato (s.l.) antibodies at screening are excluded.
* Tick bite within 3 weeks prior to screening, or tick bite during vaccination period (i.e. Day 0 to Day 56).
* Known active infection with Babesia microti (babesiosis) or Anaplasma phagocytophilum (ehrlichiosis).
* Active or passive immunization four weeks before first vaccination at Visit 1 and up to Day 84 (i.e. 4 weeks after the last VLA15 immunization). Afterwards, vaccinations should be avoided, except for influenza (seasonal or pandemic) vaccines which may be administered after Day 84 (i.e. 4 weeks after the last VLA15 immunization). Subjects susceptible to require a vaccine during the study period (e.g. due to planned travel) should be excluded at screening.
* Known congenital, hereditary or acquired immunodeficiency, including infection with human immunodeficiency virus (HIV), status post organ transplantation or immuno-suppressive therapy within 30 days prior to Day 0 and up to Day 84. Immuno-suppressive therapy is defined as administration of chronic (longer than 14 days) prednisone or equivalent ≥ 0.05 mg/kg/day. Topical and inhaled steroids are allowed.
* Planned intake of NSAID (Nonsteroidal anti-inflammatory drug) within three days prior and within seven days after any VLA15 vaccination.
* History of severe hypersensitivity reactions and anaphylaxis.
* History of allergic bronchial asthma and severe allergic rhinoconjunctivitis.
* Known hypersensitivity or allergic reactions to one of the components of the vaccine.
* History of autoimmune disease, including Type I Diabetes mellitus. Subjects with vitiligo or thyroid disease taking thyroid hormone replacement are not excluded.
* Any malignancy in the past 5 years. If treatment for cancer was successfully completed more than 5 years ago and the malignancy is considered to be cured, the subject may be enrolled.
* Acute febrile infections within 4 weeks prior to first vaccination and body temperature >37.8 C (oral) prior to each vaccination.
* Known or suspected alcohol abuse, alcohol dependence, i.e. an average of more than approximately 60 g alcohol (approximately 1 liter of beer or 0.5 liter of wine) per day] or illicit drug use within the last year;
* Inability or unwillingness to avoid more than the usual intake of alcohol (i.e. not more than 60 g alcohol (approximately 1 liter of beer or 0.5 liter of wine) per day) during the 48 hours after vaccination.
* Pregnancy (positive pregnancy test), lactation or inadequate contraception in women with childbearing potential
* Inability or unwillingness to provide informed consent or not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
* Donation of blood or blood-derived products (e.g. plasma) within 4 weeks prior to Visit 0 (Screening Visit) and during the entire study.
* Receipt of blood or blood-derived products in the past 3 months prior to Visit 0 (Screening Visit) or anticipation of such products during the entire study.
* Mental disorder as deemed clinically relevant by the investigator.
* History of Guillain-Barré-Syndrome (GBS).
* Any condition which might interfere with study objectives or that would limit the subject's ability to complete the study in the opinion of the investigator.
* Persons who are committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities).
* Persons who are in a dependent relationship with the sponsor, an investigator or other study team members, or the study center. Dependent relationships include close relatives and household members (i.e. children, partner/spouse, siblings, parents) as well as employees of the investigator or study center personnel.

Booster Extension:

* Individual stopping rule was met during the Initial Study.
* Subject has a known thrombocytopenia, bleeding disorder, or receipt of anticoagulants in the 3 weeks prior to booster vaccination contraindicating I.M. vaccination as judged by the investigator.
* Pathological findings in the symptom driven physical examination as deemed clinically relevant by the investigator or any clinically significant abnormal laboratory parameter of hematology, clinical chemistry based on investigator judgement at Visit 8. Subjects with a positive test result for RF and ACPA at Visit 8 are excluded.
* Use of any other investigational or non-registered medicinal product within 30 days prior to VLA15 booster vaccination at Visit 9 and throughout the entire Booster Extension period.
* Tick bite within 3 weeks prior to booster vaccination (i.e. Visit 9).
* Known active infection with Babesia microti (babesiosis) or Anaplasma phagocytophilum (ehrlichiosis).
* Active or passive immunization four weeks before and within 7 days after booster vaccination at Visit 9.
* Known congenital, hereditary or acquired immunodeficiency, including infection with human immunodeficiency virus (HIV), status post organ transplantation or immuno-suppressive therapy within 30 days prior to booster vaccination and up to 28 days after. Immuno-suppressive therapy is defined as administration of chronic (longer than 14 days) prednisone or equivalent ≥ 0.05 mg/kg/day. Topical and inhaled steroids are allowed.
* Developed any of the following conditions since enrolment into Initial Study:

  1. Chronic illness related to Lyme borreliosis (LB), a history of or active symptomatic LB as suspected or diagnosed by a physician.
  2. Severe cardiovascular, respiratory (including asthma), metabolic, neurological, hepatic, rheumatic, hematological, gastrointestinal, renal disorders.
  3. Musculoskeletal disorders as deemed clinically relevant by the investigator, arthritis or chronic musculoskeletal pain.
  4. Severe hypersensitivity reactions and anaphylaxis.
  5. Allergic bronchial asthma and severe allergic rhinoconjunctivitis.
  6. Hypersensitivity or allergic reactions to one of the components of the vaccine.
  7. Autoimmune disease, including Type I Diabetes mellitus. Subjects with vitiligo or thyroid disease taking thyroid hormone replacement are not excluded.
  8. Mental disorder as deemed clinically relevant by the investigator.
  9. Guillain-Barré-Syndrome (GBS)
  10. Malignancy
* Known or suspected alcohol abuse alcohol dependence, i.e. an average of more than approximately 60 g alcohol (approximately 1 liter of beer or 0.5 liter of wine per day) or illicit drug use within the last year.
* Inability or unwillingness to avoid more than the usual intake of alcohol (i.e. not more than 60 g alcohol (approximately 1 liter of beer or 0.5 liter of wine) per day) during the 48 hours after vaccination.
* Pregnancy (positive pregnancy test), lactation or inadequate contraception in women of childbearing potential.
* Inability or unwillingness to provide informed consent or not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
* Any condition which might interfere with study objectives or that would limit the subject's ability to complete the study in the opinion of the investigator.
* Persons who are committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities).
* Persons who are in a dependent relationship with the sponsor, an investigator or other study team members, or the study center. Dependent relationships include close relatives and household members (i.e. children, partner/spouse, siblings, parents) as well as employees of the investigator or study center personnel.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Rate of SAEs to Day 84 | up to Day 84 (Month 3) after first vaccination
Rate of related SAEs to Day 84 | up to Day 84 (Month 3) after first vaccination
Rate of any solicited or unsolicited Grade 3 or Grade 4 events up to Day 84 | up to Day 84 (Month 3) after first vaccination
Rate of any solicited or related unsolicited Grade 3 or Grade 4 events up to Day 84 | up to Day 84 (Month 3) after first vaccination
Rate of solicited local AEs within 7 days after each and after any vaccination up to Day 84 | up to Day 84 (Month 3) after first vaccination
Rate of solicited systemic AEs within 7 days after each and after any vaccination up to Day 84 | up to Day 84 (Month 3) after first vaccination
Rate of unsolicited AEs to Day 84, including clinically significant laboratory parameter changes | up to Day 84 (Month 3) after first vaccination
Rate of related unsolicited AEs to Day 84, including clinically significant laboratory parameter changes | up to Day 84 (Month 3) after first vaccination

SECONDARY OUTCOMES:
Rate of SAEs during the entire study period | up to Day 365 (Month 12)
Rate of related SAEs during the entire study period | up to Day 365 (Month 12)
Rate of any solicited or unsolicited Grade 3 or Grade 4 AEs during the entire study period | up to Day 365 (Month 12)
Rate of any solicited or related unsolicited Grade 3 or Grade 4 AEs during the entire study period | up to Day 365 (Month 12)
Rate of unsolicited AEs during the entire study period | up to Day 365 (Month 12)
Rate of related unsolicited AEs during the entire study period | up to Day 365 (Month 12)
Changes in laboratory parameters and rate of subjects with abnormal laboratory parameter | up to Day 365 (Month 12)
GMTs (Geometric Mean Titre) for IgG against each OspA serotype ST1 to ST6, determined by ELISA | Day 0, 28, 56, 84, 180, 236 and 365
SCRs (Seroconversion Rate, defined based on fold increase of each OspA serotype specific IgG (ST1 to ST6) as compared to baseline) | Day 28, 56, 84, 180, 236 and 365
GMFR (Geometric Mean of the fold rise as compared to baseline) for IgG against each OspA serotype ST1 to ST6, determined by ELISA | Day 28, 56, 84, 180, 236 and 365

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Pfizer CT.gov Call Center, Principal Investigator — Pfizer
Locations (5):
- United States (4):
  - eStudy Site, La Mesa, California
  - eStudySite, La Mesa, California
  - Celerion Inc., Lincoln, Nebraska
  - Celerion, Inc, Lincoln, Nebraska
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Bezay N, Hochreiter R, Kadlecek V, Wressnigg N, Larcher-Senn J, Klingler A, Dubischar K, Eder-Lingelbach S, Leroux-Roels I, Leroux-Roels G, Bender W. Safety and immunogenicity of a novel multivalent OspA-based vaccine candidate against Lyme borreliosis: a randomised, phase 1 study in healthy adults. Lancet Infect Dis. 2023 Oct;23(10):1186-1196. doi: 10.1016/S1473-3099(23)00210-4. Epub 2023 Jul 4. PMID 37419129
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=VLA15-101